CLINICAL TRIAL: NCT06666413
Title: A Single-arm, Open-label, Phase 4 Study to Evaluate the Safety and Efficacy of Avalglucosidase Alfa in Chinese Participants With Infantile-onset Pompe Disease (IOPD)
Brief Title: China Post-approval Commitment (PAC) Study of Avalglucosidase Alfa in Participants With IOPD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS18086; U1111-1295-2947 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-10-16; First posted 2024-10-30 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Glycogen Storage Disease Type II; Pompe's Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- avalglucosidase alfa (Experimental): Avalglucosidase alfa will be administered by IV infusion following reconstitution and dilution at a dose of 20 mg/kg body weight qow
  Interventions: Drug: Avalglucosidase alfa

INTERVENTIONS:
Drug: Avalglucosidase alfa — Pharmaceutical form: Sterile lyophilized powder Route of administration: IV infusion
  Other Names: GZ402666; Nexviazyme

SUMMARY:
This is a single group, 52-week treatment, Phase 4, open-label, single-arm study to assess the safety and efficacy of avalglucosidase alfa IV infusion in male and female Chinese participants with IOPD who are treatment-naïve or were previously treated with ERT.

Study details include:

* The study duration: total study duration is approximately 64 weeks.

  * Screening period of up to 8 weeks
  * Treatment period of 52 weeks
  * Follow-up period of 4 weeks.
* The number of visits will be 30, including 29 site visits and 1 phone call follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be <18 years of age, at the time of signing the informed consent.
* Participants have documented onset of Pompe disease symptoms before 12 months of age (corrected for gestation if born before 40 weeks); and diagnosis of IOPD is confirmed by GAA enzyme deficiency from any tissue source and GAA gene pathogenic mutations.
* Participants must have documented cardiomyopathy at the time of diagnosis.
* Contraceptive use should be consistent with local regulations Participant's parent/legally authorized representative (LAR) must be capable of giving signed informed consent.

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Participants with major congenital abnormality that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival.
* Participants with clinically significant organic disease (with the exception of symptoms relating to Pompe disease).
* Participants who have received an ERT other than alglucosidase alfa or avalglucosidase alfa, or any other treatment for Pompe disease, including gene therapy prior to the enrollment.
* Participants who have received alglucosidase alfa or avalglucosidase alfa less than 1 week prior to the first dose of avalglucosidase alfa given as IMP Participants who are anticipated to take prohibited therapy (ie, any other treatment for Pompe disease) during this study.
* Participants who have taken other investigational drugs (not Pompe disease specific) within 30 days or 5 elimination half-lives in blood of that drug before enrollment, whichever is longer, or are anticipated to take any other concurrent investigational treatments.
* Participants not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-05-02 (Estimated); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs, AESIs including IARs during the TE period | From baseline to Week 56
Abnormality in clinical laboratory, vital signs, and ECG parameters during the TE period | From baseline to Week 56

SECONDARY OUTCOMES:
Proportion of participants who are alive and free of invasive ventilation at Week 52 | At Week 52
Change from baseline to Week 52 in LVM Z score evaluated by echocardiography | From baseline to Week 52
The absolute change in body growth Z scores from baseline to Week 52 | From baseline to Week 52
The percentiles of the body growth Z scores changes from baseline to Week 52 | From baseline to Week 52
Change from baseline to Week 52 in distance walked during six-minute walk test (6MWT) (in applicable participants) | From baseline to Week 52
Change from baseline to Week 52 in quick motor function test (QMFT) score (in applicable participants) | From baseline to Week 52
Number of motor development milestones achieved as evaluated by Motor Milestone Checklist at Week 52 | At Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site Number: 1560001, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org